CLINICAL TRIAL: NCT06287697
Title: Determination of Energy Expenditure and Body Composition of Infants and Young Children (6-24 Months Old) in Asia Using the Doubly-Labelled Water (DLW) Technique
Brief Title: Energy Expenditure and Body Composition of Infants and Young Children (6-24 Months Old) in Asia
Status: Active, not recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: International Atomic Energy Agency (Other Government); National Institute of Nutrition, Vietnam (Other Government); Faculty of Medicine, University of Ruhuna, Sri Lanka (Unknown); Pakistan Institute of Nuclear Science and Technology (PINSTECH) (Other Government); Food and Nutrition Research Institute, Philippines (Other Government); FAO (Other)
Responsible Party: Principal Investigator, Tippawan Pongcharoen, Assistant Professor Dr., Mahidol University
Other Study IDs: LOA/RAP/2019/20
Record Dates: First submitted 2024-01-11; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Energy Expenditure; Body Composition; Infants and Young Children; Infant and Young Child Feeding
Keywords: Total energy expenditure; Fat mass; Fat-free mass; Doubly-labelled water; Children aged 6-24 months; Infant and young child feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Longitudinal study-Thailand: Cohort 1: 60 children were started at 6-8 months old, and were followed-up at 9-11, 12-14 and 15-17 months old.
  Cohort 2: 71 children were started at 12-14 months old, were followed-up 15-17, 18-21 and 21-24 months old.
  Interventions: Other: No intervention
- Cross-sectional study-Pakistan: Children aged 6-8, 9-11, 12-14, 15-17, 18-20, 21-23 months, both sexes.
  Interventions: Other: No intervention
- Cross-sectional study-Philippines: Children aged 6-8, 9-11, 12-14, 15-17, 18-20, 21-23 months, both sexes.
  Interventions: Other: No intervention
- Cross-sectional study-Sri Lanka: Children aged 6-8, 9-11, 12-14, 15-17, 18-20, 21-23 months, both sexes.
  Interventions: Other: No intervention
- Cross-sectional study-Vietnam: Children aged 6-8, 9-11, 12-14, 15-17, 18-20, 21-23 months, both sexes.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This project is a collaboration between International Atomic Energy Agency (IAEA), FAO Regional Office for Asia and The Pacific, and Mahidol University, Thailand to carry out the study on doubly-labeled water for assessment of total energy expenditure and body composition among infants and young children aged 6-23 months old. Thailand conducted a longitudinal study with participation from 4 other countries, namely, Pakistan, Philippines, Sri Lanka and Vietnam, in undertaking the same assessments in a cross-sectional design.

DETAILED DESCRIPTION:
The current international recommendations on energy requirements for children aged 6-24 months were established based on data from the Western populations. More human data of healthy children from the developing countries where the living conditions may not be as favourable for child growth and development would be needed to ascertain the validity of the global recommendation. The role of the doubly-labelled water (DLW) technique in measuring total daily energy expenditure to derive energy requirements for humans was also highlighted. Low and middle income countries in Asian countries have undergone the nutrition transition and malnutrition on both ends of the spectrum emerge as significant nutrition challenges during this critical period of growth. Unfortunately, data on body composition, i.e., the relative amounts of fat and lean or fat-free tissue which constitutes quality normal growth beyond anthropometric measurements are scarce. These data will also be needed to guide the infant and young child feeding (IYCF) recommendations for good nutrition and health and to prevent all forms of malnutrition in the region.

This project addressed the need to fill the information gap for the region, and potentially be included for making revision on energy requirement recommendations for infants and young children (IYC) for Asia and beyond. Building on the previous technical cooperation between institutions in Southeast and South Asia with the International Atomic Energy Agency (IAEA) on stable isotopic techniques for health and nutrition well-being, this project is a collaboration between IAEA, FAO Regional Office for Asia and The Pacific, and Mahidol University, Thailand to carry out the study on doubly-labeled water for assessment of total energy expenditure and body composition among infants and young children aged 6-23 months old. Thailand conducted a longitudinal study with participation from 4 other countries, namely, Pakistan, Philippines, Sri Lanka and Vietnam, in undertaking the same assessments in a cross-sectional design.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* Being aged >18 y old
* Being non-smoker
* Gestational age at delivery 37-41weeks
* Belonging to the major ethnicity of the country
* Having any socio-economic status
* Willing to sign informed written consent

Inclusion Criteria for Infants:

* Healthy baby
* Full term
* Having birth weight between 2.5 and 4.0 kg
* Height-for-age Z score and weight-for-height Z score at or above -2SD
* Being exclusively or predominantly breast-fed for at least 3 months

Exclusion Criteria for Mothers:

* Mothers: having chronic diseases, e.g., gestational diabetes were excluded.

Exclusion Criteria for Infants:

* Having inborn errors or chronic diseases e.g., celiac diseases
* Taking special supplement, e.g., RUTF.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Apparently healthy infants and young children aged 6-23 months of both sexes, belonging to the major ethnicity of the country, and having any socio-economic status.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Total Energy Expenditure | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Total Energy Expenditure assessed using doubly labelled water (DLW) technique
Body composition | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Body composition assessed using doubly labelled water (DLW) technique

SECONDARY OUTCOMES:
Weight | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Body weight of infants in kilograms
Length | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Lenght of infants in centimeters
Head circumference | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Head circumference of infants in centimeters
Mid-upper arm circumference | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Mid-upper arm circumference of the left arm in centimeters
Triceps skinfold thickness | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Triceps skinfold thickness of the left arm in millimeters
Subscapular skinfold thickness | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  Subscapular skinfold thickness of the left side in millimeters
Infant and Young Child Feeding (IYCF) | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  IYCF indicators were determined using the IYCF questionnaire IYCF practices were assessed using the IYCF , breast milk intake, dietary intake
Dietary intake | assessed at aged 6-8, 9-11, 12-14, 15-17, 18-20, and 21-23 months
  24-hr recall was administered for 3 days to obtain nutrient intakes from breast milk and diet

CONTACTS AND LOCATIONS:
Overall Officials: Tippawan Pongcharoen, PhD, Principal Investigator — Mahidol University
Locations (1):
- Institute of Nutrition, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IAEA repository upon approval
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2025 onward
Access Criteria: Upon approval

REFERENCES:
- [Result] Ua-Areechit T, Suteerojntrakool O, Pongcharoen T, Winichagoon P, Judprasong K, Murphy-Alford AJ, Lee WTK, Potip B, Sridonpai P, Tongchom W, Chomtho S. Breastfeeding duration is associated with higher adiposity at 6-8 months of age. Matern Child Nutr. 2023 Jan;19(1):e13438. doi: 10.1111/mcn.13438. Epub 2022 Oct 18. PMID 36254499